CLINICAL TRIAL: NCT01126710
Title: Optical Detection of Intravenous Infiltration
Status: Completed | Type: Observational
Sponsor: CW Optics, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Leonard Winchester, Ph.D., Chief Scientific Officer, CW Optics, Inc., CW Optics, Inc.
Other Study IDs: IV-2010-01; 5R44HL062008-06 (NIH)
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Intravenous Infiltration; Extravasation of Diagnostic and Therapeutic Materials
Keywords: infiltration; extravasation; optical monitoring
MeSH Terms: conditions — Extravasation of Diagnostic and Therapeutic Materials

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of an optical device designed and developed for monitoring the intravenous infusion site for infiltration. The hypothesis is that the changes in optical signals measured near the infusion site using the optical device can be used to monitor intravenous infusion for infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have peripheral IV catheter with active infusions that are anticipated to be in place and functioning for 48-72 hours. The IVs and accompanying infusions are solely a part of the subject's medical care and are not started or terminated for the purposes of this Study. The rationale for choosing this time frame is that the rate of infiltration is likely to be increased the longer the IV infusion is taking place.
* Subjects are admitted to one of the institution's intensive care or intermediate care units, including Adult Emergency Department, Pediatric Emergency Department, Adult Medical Intensive Care Unit, Pediatric Intensive Care Unit, Neonatal Intensive Care Unity, Surgical-Trauma Intensive Care Unit, Cardiothoracic Surgery Intensive Care Unit, Neuroscience Intensive Care Unit, Burn Intensive Care Unit, Transplant Intensive Care Unit, Coronary Care Intensive Care Unit, Post-Anesthesia Recovery Unit, Pediatric Intermediate Care Unity, Surgical Intermediate Care Unit, and Medical Intermediate Care Unit.

Exclusion Criteria:

* Inability to consent
* Lack of a peripheral IV

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects recruited from the patient population at Virginia Commonwealth University Health System will be enrolled in the Study.
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2010-05

PRIMARY OUTCOMES:
Test performance of novel optical device for monitoring intravenous infusion site for infiltration. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University Health System, Richmond, Virginia, United States